CLINICAL TRIAL: NCT03215199
Title: Northern Alberta Psychosocial Telecare (NAPT) Screening for Surgical Head and Neck Cancer Patients: a Randomized Controlled Trial
Brief Title: Northern Alberta Psychosocial Telecare (NAPT) Screening for HNC Patients
Acronym: NAPT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HREBA.CC-17-0160
Record Dates: First submitted 2017-07-09; First posted 2017-07-12 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Cancer Distress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Group (No Intervention): The Usual Care Group will include adult patients undergoing primary surgical treatment for head and neck cancer. Supportive care will be offered or provided according to patients' wishes.
- NAPT Group (Active Comparator): The NAPT Group will include adult patients undergoing primary surgical treatment for head and neck cancer. Patients will be given access to a web-based application that monitors depression, distress, and functional outcomes scores at regular intervals for 12 months. Patients will be able to alert the treatment team of decreased mood, increased distress, and functional issues impacting both. Patients will also be able to track their mood and distress levels throughout the 12 months and involve care-givers in monitoring as well.
  Interventions: Other: NAPT

INTERVENTIONS:
Other: NAPT — Web-based depression and distress monitoring application
  Arms: NAPT Group

SUMMARY:
This is a randomized controlled trial comparing a web-based psychosocial screening application to usual care in a cohort of surgically-treated head and neck cancer patients to determine its efficacy in monitoring depression and distress, and prompting necessary psychiatry/psychology referrals. In addition, treatment adherence, rehabilitation and return to work, primary care utilization, and survival will be monitored.

DETAILED DESCRIPTION:
This is a randomized controlled trial comparing a web-based psychosocial screening application to usual care in a cohort of surgically-treated head and neck cancer patients.

This study will utilize a web-based application available on desktop or laptop computers, and smartphones. The application involves monitoring using the NCCN Distress Thermometer Score, the Quick Inventory of Depressive Symptomatology-Self Report (QIDS-SR) score, and the Head and Neck Research Network (HNRN-33), a patient-reported, validated functional outcomes score. These assessments will be completed at baseline, 2 weeks postoperatively, and monthly thereafter until 12 months. Patients will have the option of filling out questionnaires more frequently if desired.

This web-based application, the NAPT App, will allow patients to alert the treatment team of their current state of mood or distress. Automatic alerts will be sent to the team if a Distress Score of </=3, a QIDS score >/=11, or suicidal ideation are expressed in the application.

The study duration will be 12 months with a primary endpoint of 6 months. Our primary outcome will be NCCN Distress Thermometer Score at 6 months, with secondary outcomes of the QIDS and HNRN-33 functional scores at 6 and 12 months. Additional outcomes assessed will pertain to completion of adjuvant therapy, weight maintenance, rehabilitation and return to work, and survival. Health services delivery outcomes, such as primary care visits, emergency department visits, hospitalizations, and narcotic use will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 18 years
* New (non-recurrent) head and neck cancer
* Primary surgical treatment

Exclusion Criteria:

* <18 years
* Recurrent head and neck cancer
* Previous chemotherapy or radiation therapy
* History of psychiatric or psychologic illness
* History of previous cancers or cancer distress

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Distress Thermometer Score | 6 months
  NCCN Distress Thermometer Score

SECONDARY OUTCOMES:
QIDS Score | 6 and 12 months
  Quick Inventory of Depressive Symptomatology-Self Report (QIDS-SR)
HNRN-33 | 6 and 12 months
  Head and Neck Research Network (HNRN-33)
Completion of Adjuvant Therapy | 6 months
  Completion of Adjuvant Therapy, including radiation or chemotherapy
Return to work | 12 months
  Return to work by 12 months
Hospital Readmissions | 12 months
  Hospital Readmissions
Primary Care Visits | 12 months
  Primary Care Visits to Family Physician
Emergency Department Visits | 12 months
  Emergency Department Visits

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No